CLINICAL TRIAL: NCT03139630
Title: COPANA - A09 PCSK 9 Substudy: Impact of Protease Inhibitors on PCSK9 Levels in Naive HIV-Infected Patients
Acronym: COPANA
Status: Completed | Type: Observational
Sponsor: Franck Boccara (Other)
Collaborators: National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Amgen (Industry)
Responsible Party: Sponsor-Investigator, Franck Boccara, Professor, Senior Cardiologist, Deputy Director of the Division of Cardiology, Saint Antoine University Hospital
Organization: Saint Antoine University Hospital (Other)
Other Study IDs: COPANA - A09 PCSK 9 substudy
Record Dates: First submitted 2016-12-26; First posted 2017-05-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: HIV Seropositivity; Dyslipidemias; PCSK9
Keywords: HIV, Dyslipidemia; Dyslipidemia; Protease Inhibitor; Ritonavir; PCSK9; Observational
MeSH Terms: conditions — HIV Seropositivity; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples taken from the Biobank stored at Tenon Hospital, Paris (Biochemistry department).
  ELISA Cyclex.
  Plasma PCSK9 concentrations assayed in triplicates using a quantitative sandwich ELISA assay and following the manufacturer instructions (Circulex CY-8079, CycLex Co, Nagano, Japan).
  The ELISA kit relies on a quantitative sandwich enzyme immunoassay technique with inter- and intraplate CVs of 2.9-7.3% and 1.5-2.6%, respectively.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-infected patients: HIV-infected adult male or female patients who are HIV treatment naive and initiate antiretroviral therapy including a protease inhibitor during the follow up period.
- HIV-uninfected patients: HIV-uninfected adult male or female patients.

SUMMARY:
Evaluation of the impact of initiation of protease inhibitor/ritonavir on PCSK9 levels in HIV-infected antiretroviral-naïve patients from the ANRS C09 COPANA cohort.

DETAILED DESCRIPTION:
Background: HIV-infected subjects are at high risk of coronary heart disease (CHD) partly in relation with atherogenic dyslipidemia including increased triglycerides (TG) and LDL-cholesterol (LDL-C). Mechanisms of HIV-associated dyslipidemia are complex, involving HIV itself and some antiretrovirals (ARV), particularly protease inhibitors (PI/r). Elevated proprotein convertase subtilisin kexin 9 (PCSK9) level is associated with increased LDL-C in the general population. How PCSK9 level is regulated in HIV-infected treated patients has never been investigated.

Objectives: We aimed to identify factors associated with circulating PCSK9 concentration in ART-naïve and treated patients and to evaluate the impact of 1st line ARV therapy (ART) comprising a PI/r, on PCSK9 level in HIV-infected patients.

Methods: Fasting plasma concentrations of PCSK9 were measured using ELISA assay in HIV-infected individuals from the ANRS COPANA cohort, at ART initiation and after one year of PI/r-based therapy without any disruption. Subjects not virologically suppressed at follow-up, or taking any lipid lowering therapies at baseline or during follow-up were excluded. Spearman's correlation coefficient was used to determine the association between PCSK9 levels and metabolic parameters at baseline and under PI/r.

ELIGIBILITY:
Inclusion Criteria:

* Naive HIV-infected male or female > 18 years
* Initiation of antiretroviral therapy including a protestase inhibitor during the follow up with blood samples available
* Patients controlled at one year with a VL<400 copies/ml

Exclusion Criteria:

* Subjects under statin or other lipid lowering drugs (fenofibrate, ezetimibe)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients: adult male or female patients who are HIV treatment naive and initiate antiretroviral therapy including a protease inhibitor during the follow up period.
  HIV-uninfected patients: adult adult male or female patients.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
PCSK9 plasma level change after initiation of ART including protease inhibitor boosted with ritonavir (PI/r) | 1 year
  Mean percent change in PCSK9 plasma levels after initiation of ART including protease inhibitor boosted with ritonavir (PI/r)r in naïve HIV-infected patients: comparison of values at ART initiation.

SECONDARY OUTCOMES:
PCSK9 correlation with lipid parameters | 1 year
  Correlations between PCSK9 levels under PI/r and lipid parameters (LDLc, HDLc, triglycerides) and other parameters (glycemia, HOMA_IR) - from baseline to end.
PCSK9 correlation with inflammatory makers/adipocytokines | 1 year
  Comparison of inflammatory makers/adipocytokines (IL6, hsCRP, leptin, adiponectin) and PCSK9 change - from baseline (naive) to after ART initiation.
PCSK9 comparison between HIV-infected and uninfected patients | 1 year
  Comparisons of PCSK9 levels between controls (HIV-uninfected from blood donors) and HIV-infected patients - from baseline (naive) and after ART initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Boccara, MD, PhD, Principal Investigator — Saint Antoine University Hospital
Locations (1):
- Cardiology Department, Saint Antoine University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Derived] Boccara F, Ghislain M, Meyer L, Goujard C, Le May C, Vigouroux C, Bastard JP, Fellahi S, Capeau J, Cohen A, Cariou B; ANRS-COPANA Study Group. Impact of protease inhibitors on circulating PCSK9 levels in HIV-infected antiretroviral-naive patients from an ongoing prospective cohort. AIDS. 2017 Nov 13;31(17):2367-2376. doi: 10.1097/QAD.0000000000001633. PMID 28857822